CLINICAL TRIAL: NCT07073079
Title: Second-line Advanced Therapy in Crohn's Disease: Real-life Effectiveness and Resolution of First-line Suboptimal Control Indicators (CROHNOS - CROHN Therapy Observational Study)
Brief Title: A Study to Assess the Effectiveness of Second-Line Therapy of Upadacitinib and Risankizumab in Adult Participants With Crohn's Disease in a Real-World Setting
Acronym: CROHNOS
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P25-397
Record Dates: First submitted 2025-06-02; First posted 2025-07-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Upadacitinib; Risankizumab
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Upadacitinib: Participants with Crohn's Disease prescribed upadacitinib in routine clinical practice are observed from the first dose up to 18 months.
- Risankizumab: Participants with Crohn's Disease prescribed risankizumab in routine clinical practice are observed from the first dose up to 18 months.

SUMMARY:
Crohn's disease (CD) is an incurable chronic inflammatory disorder of the gastrointestinal tract. This study will evaluate the second line effectiveness of upadacitinib and risankizumab in Crohn's Disease (CD) in a real-world setting.

Upadacitinib and risankizumab are approved drugs for treating CD. Approximately 250 participants who are prescribed upadacitinib or risankizumab by their physician in accordance with local label will be enrolled in 25 sites across Italy.

Participants will receive upadacitinib or risankizumab as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed for up to 18 months.

No additional burden for participants in this trial is expected.

DETAILED DESCRIPTION:
The retrospective phase will be up to 2 years prior to enrollment to the study, the prospective phase will be up to 18 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of moderate-to-severe Crohn's Disease (CD) confirmed by clinical, and/or endoscopic/histological indexes
* Participants previously treated with Tumor Necrosis Factor inhibitor (TNF-i) as fist line (1L) therapy for at least 6 months; clinical documentation available in medical charts for the previous 2 years or since the beginning of the 1L therapy

Exclusion Criteria:

* Any condition included in the "warning and precautions" and "contraindications" section of the approved local upadacitinib/risankizumab label
* Participants previously exposed to upadacitinib/risankizumab or any approved or investigational non TNFi biologic Disease Modifying Antirheumatic Drug (bDMARDs) for CD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with Crohn's Disease
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve Corticosteroids (CS) Free Remission | Month 12
  CS free remission is defined as clinical remission with Harvey Bradshaw Index (HBI) <4 and absence of corticosteroid use since at least three months prior to month 12.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (23):
- Italy (23):
  - Ospedale Specializzato In Gastroenterologia Saverio De Bellis /ID# 275706, Castellana Grotte, Bari
  - Azienda Ospedaliero Universitaria di Cagliari - P.O. Duilio Casula /ID# 275216, Monserrato, Cagliari
  - Fondazione di Religione e di Culto Casa Sollievo della Sofferenza /ID# 275669, San Giovanni Rotondo, Foggia
  - Ospedale San Martino /ID# 274529, Genoa, Genova
  - IRCCS Istituto Clinico Humanitas /ID# 274489, Rozzano, Lombardy
  - IRCCS Ospedale San Raffaele /ID# 274458, Milan, Milano
  - Fondazione IRCCS San Gerardo dei Tintori - Ospedale San Gerardo /ID# 274682, Monza, Monza E Brianza
  - Azienda Ospedaliera Universitaria Federico II /ID# 274570, Naples, Napoli
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli /ID# 274788, Naples, Napoli
  - A.O.U. CITTA' DELLA SALUTE E DELLA SCIENZA DI TORINO - Ospedale Molinette /ID# 274461, Turin, Piedmont
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 274654, Rome, Roma
  - Ospedale Sandro Pertini /ID# 275023, Rome, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Universita Cattolica /ID# 274530, Rome, Roma
  - A.O. Ordine Mauriziano di Torino /ID# 274459, Turin, Torino
  - IRCCS Ospedale Sacro Cuore Don Calabria /ID# 274462, Negrar, Verona
  - A.O.U. Consorziale Policlinico di Bari /ID# 274662, Bari
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 275161, Bologna
  - AOU Policlinico G. Rodolico - San Marco /ID# 274909, Catania
  - Azienda Ospedaliera di Catanzaro Pugliese Ciaccio /ID# 274571, Catanzaro
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico /ID# 274618, Milan
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello /ID# 274964, Palermo
  - Fondazione Policlinico Universitario Campus Bio-Medico /ID# 274488, Roma
  - Fatebenefratelli Isola Tiberina - Gemelli Isola /ID# 274966, Roma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P25-397